CLINICAL TRIAL: NCT02842619
Title: Phase I/II Open Label First in Human Single Center Clinical Study Aimed to Evaluate the Safety and Efficacy of BonoFill-II in Reconstructing Maxillofacial Bone
Brief Title: Filling Bone Defects/Voids With Autologous BonoFill-II for Maxillofacial Bone Regeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BonusBio Group Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CP-BNS03
Record Dates: First submitted 2015-11-24; First posted 2016-07-25 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Bone Augmentation; Bone Grafts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention Arm (Experimental): 1 Arm - IMP treatment arm
  Interventions: Biological: BonoFill-II

INTERVENTIONS:
Biological: BonoFill-II — Sinus augmentation - Surgery will be performed by either open or close sinus augmentation as per investigator discretion and as per common medical practice. After the elevation, BonoFill-II will be transplanted on the residual sub-antral bone.
  Bone grafting after removal of cysts from jaws - Treatment will be performed according to the size of the cyst: in relatively small cyst total enucleation will be performed. In large cysts, a process of marsupialization will be performed. The entire cyst will be removed, including the epithelium layer, and the BonoFill-II product will be used for filling.

SUMMARY:
The purpose of this clinical study is to evaluate the safety and the efficacy of BonoFill-II as a bone filler containing the patient's own (autologous) adipose (fat) tissue-derived cells in reconstructing bone in two clinical indications:

1. Bone augmentation (e.g. sinus augmentation)
2. Bone grafting after removal of cysts from jaws

DETAILED DESCRIPTION:
Safety endpoint:

The transplantation of BonoFill-II to the maxillary or mandible defect/void is safe under the following conditions: No chronic bone infection (Osteomyelitis); no significant changes in complete blood count (CBC) and in general health.

Efficacy endpoint:

The transplantation of BonoFill-II to the maxillary or mandible void is efficient: the bone defects/voids are filled with at least 8mm of total bone height at the transplanted area.

ELIGIBILITY:
Inclusion Criteria:

GENERAL

1. Subject in general good health in the opinion of the investigator as determined by medical history, vital signs physical examination and safety lab tests
2. Subject has a rehabilitation dentist and rehabilitation program
3. Up to date panoramic X-Ray/CT
4. Subject has provided written informed consent to participate in the study, understands all study procedures and agrees to follow up procedures
5. Subject is in good oral hygiene condition as per investigator's discretion

SINUS AUGMENTATION

1. The subjects requires sinus augmentation as per investigator's discretion
2. Healthy condition of Maxillary Sinuses and Oral Mucosa determined by X-ray

BONE GRAFTING AFTER REMOVAL OF CYSTS FROM JAWS

1. Subject who according to investigator diagnosis required removal of cysts from jaws. Limited to cysts diagnosed as: radicular cysts, residual cysts, congenital cysts, developmental and acquired cysts.
2. Subject's cyst was removed after diagnosis of the cyst type

Exclusion Criteria:

1. Subject with a recorded medical history of diseases such as diabetes mellitus, heart diseases, renal failure, osteoporosis, Multiple sclerosis,
2. Subject treated with systemic steroids
3. Subject with a known autoimmune disease, such as Addison's disease, Myasthenia gravis, Pernicious anemia, Reactive arthritis, Rheumatoid arthritis, Sjogren syndrome, Systemic lupus erythematosus, Type I diabetes.
4. Subject has vitiligo or a known scar healing problems (keloid formation)
5. Subject treated with Oral Bisphosphonate drugs (such as Fosalan and other similar medications)
6. Subjects underwent one of the following treatments up to 12 months prior to Visit 1: Chemotherapy, Radiotherqapy
7. In case of sinus augmentation - unhealthy conditions of Maxillary Sinuses.
8. Subject with current active infection or illness.
9. Subject participating in another clinical trial 30 days prior to and during the study period.
10. Subject is a pregnant or lactating woman. Pregnancy will be verified by urine test during screening.
11. Subject has a known history of any significant medical disorder, which in the investigator's discretion contraindicates the subject's participation.
12. Subject has a known allergy for anesthesia.
13. Subjects with known allergy to hyaluronic acid.
14. Subjects with known allergy to HypoThermosol® or Dextran-40.
15. Subjects with known allergy to any of the antibiotics: Bacitracin, Gentamicin and/or Polymyxin B Sulfate.
16. Positive serology for either HIV, hepatitis B or hepatitis C.
17. Abnormal clinically significant laboratory test and exams findings as per investigator's discretion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07-23 (Actual); Primary Completion 2024-06-02 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Safety of Bonofill-ll Administration | 6-month clinical Follow Up
  The study will assess the safety of the BonoFill-II drug product post transplantation by demonstrating No chronic bone infection (Osteomyelitis); no significant changes in complete blood count (CBC) and in general health.
Efficacy of Bonofill-ll Administration | 6-month clinical Follow Up
  Following BonoFill-II transplantation, the bone regeneration in the operated site will be evaluated using CT or panoramic X Ray. Bone formation at the implantation site inside the maxillary sinus will be evaluated by measuring the bone height at the end of the study (residual + Augmented bone at 3 evenly-spaced locations). Successful bone regeneration is achieved if:
  * Bone formation inside the maxillary sinus or bone void, in the area of dental implantation defined at Visit 1 (prior to BonoFill-ll transplantation), with average height (residual + augmented bone) of at least 8mm, OR
  * Bone formation inside the maxillary sinus in the area of dental implantation defined at Visit 1 (prior to BonoFill-II transplantation), allowing successful dental implantation.

CONTACTS AND LOCATIONS:
Overall Officials: Vered Kivity, PhD, MBA, Study Director — Bonus BioGroup
Locations (1):
- Oral and Maxillofacial Surgery Clinic - Beit Merik, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No